CLINICAL TRIAL: NCT00366587
Title: Contralateral Eye Comparison of Visual Outcomes and Patient Satisfaction After Routine Phacoemulsification and Implantation of ReSTOR and ReZoom IOLs
Brief Title: Comparison of Visual Outcomes and Patient Satisfaction After Cataract Surgery and Implantation of ReSTOR and ReZoom IOLs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MRC-06-004
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2006-07

CONDITIONS: Cataract Extraction
MeSH Terms: interventions — Cataract Extraction

INTERVENTIONS:
Device: Cataract surgery and IOL implantation

SUMMARY:
Cataract is prevalent throughout the world and IOLs are routinely implanted after the extraction of the cataractous lens. It is the most frequently performed surgery in the United States with an estimated 2-3 million procedures performed annually. With the aging population on the rise, as well as the increasing popularity of refractive intraocular lenses, the number of intraocular surgeries continues to rise. Over the years, the surgical technique has evolved from intracapsular extraction to modern phacoemulsification. This development has helped with the evolution of IOLs as well. The IOLs have advanced extensively: different materials and designs are available, permitting implantation through smaller, sutureless incisions. Traditional IOLs are of monofocal design providing vision at one distance, typically far. Patients implanted with traditional monofocal IOLs usually require glasses for near distance tasks such as reading. The new multifocal IOLs offer the possibility of seeing well at more than one distance, without glasses or contacts.

The AcrySof ReSTOR (Alcon Laboratories) uses apodized diffractive technology - a design that responds to how wide or small the eye's pupil might be - to provide near, intermediate, and distance vision. Clinical studies used to support the March 2005 FDA approval showed that 80% of people who received the lens did not use glasses for any activities after their cataract surgery; 84% who received the lens in both eyes had distance vision of 20/25 or better, with near vision of 20/32 or better.

ReZoom (Advanced Medical Optics) is a multifocal refractive zonal IOL that distributes light over five optical zones to provide near, intermediate, and distance vision. The ReZoom is a second-generation multifocal and was FDA-approved in March 2005. In a European study of 215 patients, 93% of ReZoom recipients reported never or only occasionally needing glasses. The combined use of multifocal intraocular lenses is often a solution to best meet the patients' refractive needs. There has been speculation that the implantation of ReSTOR in one eye and ReZoom lens in the fellow eye can provide patients a larger range of useful vision in the near range.

The purpose of this study is to evaluate visual outcome and patient satisfaction after implantation of a diffractive multifocal IOL (ReSTOR) in one eye and a refractive multifocal IOL (ReZoom) in the fellow eye after routine phacoemulsification and compare it to a control group of patients implanted bilaterally with ReSTOR with both eyes targeted for 0 to ±0.25 D, and to a group of patients implanted bilaterally with ReSTOR with the non-dominant eye targeted for +1.00 D and the dominant eye targeted for 0 to +0.25 D.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have an age-related cataract in both eyes.
* 18 years of age or older.
* Patient must desire cataract extraction.
* Expected maximum of 4 weeks and minimum of 1 week interval between first and second eye surgeries.
* Willing and able to comply with scheduled visits and other study procedures.

Exclusion Criteria:

* Preoperative ocular pathology: amblyopia, rubella cataract, proliferative diabetic retinopathy, shallow anterior chamber, macular edema, retinal detachment, aniridia or iris atrophy, uveitis, history of iritis, iris neovascularization, medically uncontrolled glaucoma, microphtalmus or macrophtalmus, optic nerve atrophy, macular degeneration (with anticipated best postoperative visual acuity less than 20/30), advanced glaucomatous damage, etc.
* Keratometric astigmatism exceeding 2.0 diopters.
* Planned postoperative refraction for mono-vision.
* Uncontrolled diabetes.
* Use of any systemic or topical drug known to interfere with visual performance.
* Contact lens use during the active treatment portion of the trial.
* Any concurrent infectious/non infectious conjunctivitis, keratitis or uveitis.
* Pregnant or nursing mothers and females of childbearing potential not practicing a reliable and medically acceptable method of birth control.
* Any clinically significant, serious or severe medical or psychiatric condition that may increase the risk associated with study participation or study device implantation or may interfere with the interpretation of study results.
* Participation in (or current participation) any investigational drug or device trial within the previous 30 days prior to the start date of this trial.
* Intraocular conventional surgery within the past three months or intraocular laser surgery within one month in the operated eye.
* Other ocular surgery at the time of the cataract extraction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2006-02; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Solomon, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Storm Eye Institute, Medical University of South Carolina, Charleston, South Carolina, United States